CLINICAL TRIAL: NCT04205201
Title: The Effectiveness of Topical Latanoprost Compared With Topical Brimonidine in the Treatment of the Primary Open Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chittagong Medical College (Other)
Responsible Party: Principal Investigator, Abul Khayer, Student, Chittagong Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMC/PG/2018/1828
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: To See the Safety and Efficacy of the Topical Latanoprost Compared With Topical Brimonidine in the Treatment of the Primary Open Angle Glaucoma Patients
MeSH Terms: interventions — Drugs, Investigational; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Generated by pharmaceutical companies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Latanoprost
  Interventions: Drug: Drugs, Investigational
- Group B (Other): Brimonidine
  Interventions: Drug: Drugs, Investigational

INTERVENTIONS:
Drug: Drugs, Investigational — To see the safety and efficacy of topical latanoprost compared with topical brimonidine in the treatment of the primary open angle
  Other Names: Brimonidine

SUMMARY:
Outpatient department of cmch, ceitc,cimch POAG patients enrolled for the study.

ELIGIBILITY:
Inclusion Criteria:

* IOP 22_34mmof Hg,newly diagnosed case, bilateral POAG patients Patients.

Exclusion Criteria:

* pregnant and lactating women, infection, any eye surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18_90years
Enrollment: 80 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
More than 20% IOP reduction | 0_3 months
  From baseline to month 3

SECONDARY OUTCOMES:
Adverse reaction | O_3 months
  Record every follow up period baseline to month 3.

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - Facuity of basic science and para clinical science, Dhaka, Chittagong
  - Facuity of basic scienceand para clinican science, Chittagong, Chokhbazar

IPD SHARING:
Plan to Share IPD: No